CLINICAL TRIAL: NCT02698007
Title: Safety and Benefits of Using Laryngeal Mask Airway to Keep Airway Potency During Fiber-optic Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0690-15-RMC
Record Dates: First submitted 2016-02-04; First posted 2016-03-03 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Disease Undergoing Elective Bronchoscopy.; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- without lma (No Intervention): standard fiberoptic bronchoscopy without lma
- with lma (Experimental): fiberoptic bronchoscopy with the use of lma
  Interventions: Device: Laryngeal Mask Airway (LMA)

INTERVENTIONS:
Device: Laryngeal Mask Airway (LMA) — Fiberoptic bronchoscopy with the use of LMA
  Arms: with lma

SUMMARY:
Bronchoscopy is a method of diagnosis and treatment of common respiratory diseases and lung recognized for many years.

Since the action takes place in the airways and in light of the use of sedation, when performing, the procedure requires caution to keep potent airway and breathing sufficient enough.

Most of the bronchoscopy done without the aid of equipment for advanced airway protection. During the operation done monitoring hemodynamics: such as blood pressure, pulse and respiratory such as percutaneous oxygen saturation and carbon dioxide.

Laryngeal Mask Airway (LMA) - is a tool that has been shown to be effective in securing of airway respiratory activity during positive-pressure ventilation.

Several studies have shown that the use of LMA is a convenient and safe while performing bronchoscopy for airways and lungs. However, most of the studies were for certain patient groups such as children, immuno-compromised patients.

Or benefits and safety LMA in front of intubation during bronchoscopy.

Our aim to assess the safety and efficacy LMA in not mechanically ventilated patients undergoing flexible elective bronchoscopy .

Another objective, to examine whether there is a special group of patients enjoy the LMA more than others.

Patients will be divided randomly into two groups alternately by order, one patient study group and the next one to control.

Study group : LMA is inserted under sedation and used during the procedure.

Control group - performing bronchoscopy under sedation without LMA.

About 50 people are needed each group.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 y.o
* Competency to sign informed consent.
* Room air oxygen saturation above 95%
* Stable hemodynamically and respiratory during the start procedure.
* Undergoing elective bronchoscopy.

Exclusion Criteria:

* Pregnant women and special groups will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
pulse oximetry <90%, | during bronchoscopy procedure
Percutaneous Carbon Dioxide >55%, | during bronchoscopy procedure
arrhythmia by ecg monitoring. | during bronchoscopy procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Institute,Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided